CLINICAL TRIAL: NCT03363334
Title: Expanded Access (Compassionate Use) of Fostamatinib in Patients With Persistent or Chronic Relapsing/Refractory Immune Thrombocytopenic Purpura (ITP)
Brief Title: Expanded Access of Fostamatinib in Patients With Persistent or Chronic Relapsing/Refractory ITP
Status: No longer available | Type: Expanded Access
Sponsor: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: C-935788-055
Record Dates: First submitted 2017-11-28; First posted 2017-12-06 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-06

CONDITIONS: Immune Thrombocytopenic Purpura
Keywords: ITP; Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — fostamatinib

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Fostamatinib disodium 100 mg — Fostamatinib Disodium tablet 100 mg PO bid (morning and evening)
  Other Names: Fostamatinib; R935788; R788
Drug: Fostamatinib disodium 150 mg — Fostamatinib Disodium tablet 150 mg PO bid (morning and evening)
  Other Names: Fostamatinib; R935788; R788

SUMMARY:
C-935788-055 is an open-label, multi-center, expanded access (EAP) study.

DETAILED DESCRIPTION:
The purpose of the program is to provide Fostamatinib in an Expanded Access setting to subjects who meet the selection criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient with chronic or persistent ITP.
2. Must have failed or are unable to receive standard of care treatments for ITP.
3. Must have at least two platelet counts < 30,000/µL during the last 2 months prior to screen date.

Exclusion Criteria:

1. ITP associated with lymphoma, chronic lymphocytic leukemia, transplant, or thrombocytopenia associated with myeloid dysplasia.
2. Subject has uncontrolled or poorly controlled hypertension.
3. Any of the following laboratory abnormalities: neutrophil count of < 1,500/µL, or transaminase levels (ALT, AST) > 1.5x ULN, total bilirubin > 2.0 mg/dL.
4. Active HBV or HCV infection.
5. Current or recent enrollment in an investigational drug or device study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie Duliege, M.D., Study Director — Rigel Pharmaceuticals, Inc., Chief Medical Officer